CLINICAL TRIAL: NCT05169684
Title: A Phase 2, Open-label, Randomized Controlled Trial of BMS-986218 or BMS-986218 Plus Nivolumab in Combination With Docetaxel in Participants With Metastatic Castration-resistant Prostate Cancer
Brief Title: A Study of BMS-986218 or BMS-986218 Plus Nivolumab in Combination With Docetaxel in Participants With Metastatic Castration-resistant Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA022-009; 2021-003990-74 (EudraCT Number); U1111-1268-2566 (Registry Identifier: WHO)
Record Dates: First submitted 2021-12-10; First posted 2021-12-27 (Actual); Results first posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Prostatic Neoplasms, Castration-Resistant
Keywords: BMS-986218; BMS-936558; Docetaxel; Metastatic; MDX1106; Nivolumab; ONO-4538; TAXOTERE
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant; Neoplasm Metastasis | interventions — Docetaxel; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm 1A: Docetaxel + BMS-986218 (Experimental)
  Interventions: Biological: BMS-986218; Drug: Docetaxel
- Arm 1B: Docetaxel + BMS-986218 + Nivolumab (Experimental)
  Interventions: Biological: BMS-986218; Drug: Docetaxel; Biological: Nivolumab
- Arm 2A: Docetaxel (Experimental)
  Interventions: Drug: Docetaxel
- Arm 2B: Docetaxel + BMS-986218 (Experimental)
  Interventions: Biological: BMS-986218; Drug: Docetaxel
- Arm 2C: Docetaxel + BMS-986218 + Nivolumab (Experimental)
  Interventions: Biological: BMS-986218; Drug: Docetaxel; Biological: Nivolumab
- Arm 2D (Optional Crossover): BMS-986218 + Nivolumab (Experimental)
  Interventions: Biological: BMS-986218; Biological: Nivolumab

INTERVENTIONS:
Biological: BMS-986218 — Specified dose on specified days
  Arms: Arm 1A: Docetaxel + BMS-986218; Arm 1B: Docetaxel + BMS-986218 + Nivolumab; Arm 2B: Docetaxel + BMS-986218; Arm 2C: Docetaxel + BMS-986218 + Nivolumab; Arm 2D (Optional Crossover): BMS-986218 + Nivolumab
Drug: Docetaxel — Specified dose on specified days
  Other Names: TAXOTERE
  Arms: Arm 1A: Docetaxel + BMS-986218; Arm 1B: Docetaxel + BMS-986218 + Nivolumab; Arm 2A: Docetaxel; Arm 2B: Docetaxel + BMS-986218; Arm 2C: Docetaxel + BMS-986218 + Nivolumab
Biological: Nivolumab — Specified dose on specified days
  Other Names: BMS-936558, MDX1106, ONO-4538
  Arms: Arm 1B: Docetaxel + BMS-986218 + Nivolumab; Arm 2C: Docetaxel + BMS-986218 + Nivolumab; Arm 2D (Optional Crossover): BMS-986218 + Nivolumab

SUMMARY:
The purpose of this study is to assess the safety, efficacy, tolerability, and toxicity of docetaxel alone, in combination with BMS-986218, or in combination with nivolumab plus BMS-986218 in men who have metastatic castration-resistant prostate cancer (mCRPC) that progressed after novel antiandrogen therapy and have not received chemotherapy for mCRPC.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of carcinoma of the prostate without small cell features
* Documented prostate cancer progression by Prostate Cancer Working Group 3 (PCWG3) criteria while castrate
* Evidence of metastatic disease documented by either bone lesions on radionuclide bone scan and/or soft tissue lesions on computed tomography (CT)/magnetic resonance imaging (MRI)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
* Ongoing androgen deprivation therapy (ADT) with a gonadotropin-releasing hormone (GnRH) agonist/antagonist or bilateral orchiectomy (i.e., surgical or medical castration) confirmed by testosterone level ≤ 1.73 nmol/L (50 ng/dL) at the screening visit
* Chemotherapy-naive for metastatic castration-resistant prostate cancer (mCRPC) and have received at least one novel antiandrogen therapy (NAT)

Exclusion Criteria:

* Concurrent malignancy (present during screening) requiring treatment or history of prior malignancy active within 2 years prior to treatment assignment in Part 1 or randomization in Part 2
* Untreated central nervous system (CNS) metastases
* Leptomeningeal metastases
* Active, known or suspected autoimmune disease

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (31):
- United States (25):
  - Arizona Oncology - Tucson - Wilmot Road Location, Tucson, Arizona
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Rocky Mountain Cancer Centers - Littleton, Littleton, Colorado
  - Yale School Of Medicine, New Haven, Connecticut
  - Medical Oncology Hematology Consultants - Newark, Newark, Delaware
  - The Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Local Institution - 0004, Marietta, Georgia
  - The University of Chicago Medical Center - Duchossois Center for Advanced Medicine, Chicago, Illinois
  - University Of Iowa Hospitals And Clinics, Iowa City, Iowa
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Local Institution - 0006, New York, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Oncology Hematology Care, Inc. - Eastgate, Cincinnati, Ohio
  - Willamette Valley Cancer Institute, Eugene, Oregon
  - Texas Oncology-Beaumont Mamie McFaddin Ward Cancer Center, Beaumont, Texas
  - Texas Oncology, Bedford, Texas
  - Texas Oncology - Denton North, Denton, Texas
  - Texas Oncology, Flower Mound, Texas
  - Texas Oncology - Fort Worth Cancer Center, Fort Worth, Texas
  - The University of Texas - MD Anderson Cancer Center - Genitourinary (GU) Cancer Center, Houston, Texas
  - Texas Oncology - McKinney, McKinney, Texas
  - Texas Oncology- Tyler, Tyler, Texas
  - Local Institution - 0056, Hampton, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Local Institution - 0003, Toulouse, France
- Italy (5):
  - Local Institution - 0037, Milan, MI
  - Local Institution - 0021, Rozzano, MI
  - Local Institution - 0071, Meldola
  - Local Institution - 0016, Modena
  - Local Institution - 0029, Pozzuoli

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 10 Participants enrolled and Treated. Study terminated early after safety lead in portion (part 1).
Groups:
- Treatment 1: BMS-986218 30mg Q3W + Docetaxel 75 mg/m² Q3W
- Treatment 2: BMS-986218 50mg Q3W + Docetaxel 75 mg/m² Q3W
Period: Overall Study
Arm/Group | Treatment 1 | Treatment 2
Started | 3 | 7
Completed | 1 | 0
Not Completed | 2 | 7
Not completed — Adverse Event | 1 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Progressive Disease | 1 | 1
Not completed — Participant request to discontinue treatment | 0 | 1
Not completed — Other Reason | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment 1 | Treatment 2 | Total
Number analyzed (Participants) | 3 | 7 | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.3 (6.11) | 65.7 (9.14) | 66.5 (8.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 7 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 6 | 8
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 6 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Related Adverse Events
Description: Adverse events will presented using National Cancer Institute Common Terminology Criteria for Adverse Events version 5 (NCI CTCAE v5).
Time Frame: From first dose to 100 days follow up to last dose (Approximately 22 months)
Population: All treated Participants in part 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 3 | 7
Participants | 3 | 7

2. Primary Outcome: Number of Participants With Treatment Related Serious Adverse Events
Description: as for outcome 1
Time Frame: From first dose to 100 days follow up to last dose (Approximately 22 months)
Population: All treated Participants in part 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 3 | 7
Participants | 1 | 4

3. Primary Outcome: Number of Participants With Dose Limiting Toxicities
Description: DLTs will be defined as:
  Any treatment-related AEs for which a participant permanently discontinues a study treatment (other than daily prednisone) and that occurs during the first 2 cycles of treatment.
  Any death not clearly due to the underlying disease or extraneous causes and that occurs during the first 2 cycles of treatment Greater than or equal to Grade 2 pneumonitis lasting greater than 5 days despite appropriate medical therapy and that occurs during the first 2 cycles of treatment Any neutropenic fever as well as Grade 4 neutropenia or thrombocytopenia for > 7 days that occurs during the first 2 cycles of treatment Any treatment-related AE that delays initiation of Cycle 2 or Cycle 3 of treatment by greater than 2 consecutive weeks.
Time Frame: From first dose to 100 days follow up to last dose (Approximately 22 months)
Population: All treated Participants in part 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 3 | 7
Participants | 1 | 0

4. Primary Outcome: Number of Participants With AEs Leading to Discontinuation
Description: as for outcome 1
Time Frame: From first dose to 100 days follow up to last dose (Approximately 22 months)
Population: All treated Participants in part 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 3 | 7
Participants | 2 | 4

5. Primary Outcome: Number of Participants Who Died
Description: Number of participant deaths
Time Frame: From first dose to 100 days follow up to last dose (Approximately 22 months)
Population: All treated Participants in part 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 3 | 7
Participants | 2 | 2

6. Secondary Outcome: Prostate Specific Antigen Response Rate (PSA-RR)
Description: PSA-RR is the proportion of randomized participants with a 50% or greater decrease in PSA from baseline to any post-baseline PSA result. A second consecutive value obtained 3 or more weeks later is required to confirm the PSA response.
Time Frame: From first dose to 100 days follow up to last dose (Approximately 22 months)
Population: PSA Evaluable Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 3 | 7
Percentage of Participants
  Unconfirmed or Confirmed PSA responders | 33.3 [0.8 to 90.6] | 57.1 [18.4 to 90.1]
  Confirmed PSA responders | 33.3 [0.8 to 90.6] | 57.1 [18.4 to 90.1]

7. Secondary Outcome: Objective Response Rate
Description: Objective response rate per PCWG3 (ORR-PCWG3) is the proportion of participants who have a confirmed complete or partial best overall response (BOR) per PCWG3 among randomized participants who have measurable disease at baseline. The BOR is defined as the best response designation, as determined by the BICR, recorded between the date of randomization and the date of objectively documented radiographic progression, or last tumor measurement, whichever occurs first.
Time Frame: From first dose to 100 days follow up to last dose (Approximately 22 months)
Population: Study was terminated after safety lead in portion of part 1. Efficacy Data in part 2 was not collected, which includes this endpoint.
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Time to Response
Description: Time to response per PCWG3 (TTR-PCWG3) is the time from randomization date to the date of the first documented CR or PR per PCWG3, as determined by BICR.
Time Frame: From first dose to 100 days follow up to last dose (Approximately 22 months)
Population: as for outcome 7
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Duration of Response
Description: Duration of response per PCWG3 (DOR-PCWG3) is the time between the date of first response (CR/PR per PCWG3) to the date of first documented radiographic progression per PCWG3 (as determined by BICR), or death due to any cause.
Time Frame: From first dose to 100 days follow up to last dose (Approximately 22 months)
Population: as for outcome 7
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Overall Survival
Description: OS for all randomized participants is the time between randomization date and the date of death from any cause.
Time Frame: From first dose to 100 days follow up to last dose (Approximately 22 months)
Population: as for outcome 7
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events: (From first dose to last dose + 100 days): Approximately 22 Months All-Cause mortality (From randomization to end of study): Approximately 22 Months.
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Arm/Group | Treatment 1 | Treatment 2
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/7
Serious Adverse Events (participants affected / at risk) | 1/3 | 6/7
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1 (N=3) | Treatment 2 (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 1
Vasculitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1 (N=3) | Treatment 2 (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 | 4
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Eye disorder (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Bowel movement irregularity (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 4
Constipation (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 4
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 5
Oral pain (Gastrointestinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 3
Asthenia (General disorders) | 1 | 1
Chills (General disorders) | 0 | 1
Face oedema (General disorders) | 0 | 1
Fatigue (General disorders) | 3 | 4
Generalised oedema (General disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 1
Injection site reaction (General disorders) | 0 | 1
Localised oedema (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 1
Mucosal inflammation (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 3
Pyrexia (General disorders) | 0 | 4
Swelling face (General disorders) | 0 | 1
Terminal agitation (General disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1
Candida infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Staphylococcal skin infection (Infections and infestations) | 0 | 1
Submandibular abscess (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 2
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0
Influenza A virus test positive (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1
Mycobacterium tuberculosis complex test positive (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 2
Nitrite urine present (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 2 | 1
Prostatic specific antigen increased (Investigations) | 1 | 0
Weight increased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Sacral pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 3
Dysgeusia (Nervous system disorders) | 1 | 3
Headache (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 2
Presyncope (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Cystitis noninfective (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Urethral pain (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 3
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Flushing (Vascular disorders) | 0 | 1
Hot flush (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 0 | 5
Orthostatic hypotension (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This study was terminated early after the safety lead-in portion (Part 1).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT05169684/Prot_SAP_000.pdf